CLINICAL TRIAL: NCT01471353
Title: Sorafenib Plus Capecitabine (SorCape) in Previously Treated Metastatic Colorectal Cancer
Acronym: SorCape
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC2010-23; IRB201701484 (Other: University of Florida conversion#)
Record Dates: First submitted 2011-11-10; First posted 2011-11-16 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Metastatic; Colon Cancer; Rectal Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Sorafenib; Capecitabine; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sorafenib Plus Capecitabine (SorCape) (Experimental): Sorafenib 200-400 mg PO twice daily on days 1-21 (dose escalation schema) plus Capecitabine 1000 mg/m2 PO twice daily on days 1-14 repeated every 21 days. Single arm study.
  Interventions: Drug: Sorafenib Plus Capecitabine (SorCape)

INTERVENTIONS:
Drug: Sorafenib Plus Capecitabine (SorCape) — Sorafenib 200-400 mg PO twice daily on days 1-21 (dose escalation schema) plus Capecitabine 1000 mg/m2 PO twice daily on days 1-14 repeated every 21 days
  Other Names: Nexavar; Xeloda; Chemotherapy

SUMMARY:
Combining Sorafenib with standard cytotoxic fluoropyrimidine therapy for advanced colorectal cancer may provide clinical benefit when no other treatment remains.

DETAILED DESCRIPTION:
The Raf/MEK/ERK pathway is an important mediator of responses to growth factors, and a strong inducer of genes involved in tumorigenesis, angiogenesis, apoptosis, and tumorigenesis in metastatic colorectal cancer (mCRC). Inhibition of this pathway has been previously proven to be highly clinically beneficial for patients with this disease. It has also been clearly demonstrated that the inhibition of VEGF, when coupled with cytotoxic therapy and/or continued beyond initial response, can improve clinical outcomes and survival in this same cohort of patients. Safety and pharmacokinetic data have already been established for this novel doublet oral chemotherapy. This study is intended to determine the activity of a combination of oral fluoropyrimidine plus sorafenib in an advanced mCRC patient population for whom limited treatment options remain.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven adenocarcinoma of the colon or rectum.
* Metastatic disease that is not amenable to potentially curative treatment.
* Measurable disease (as per RECIST 1.1 criteria).
* At least one prior chemotherapeutic regimen for metastatic disease. Patients must have progressed following oxaliplatin based therapy (in either the adjuvant or metastatic setting) and irinotecan based therapy (in the metastatic setting).
* Adequate bone marrow, liver and renal function.
* Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate, provided stability in anticoagulation therapy is documented at the treating provider's discretion. For patients on warfarin, the INR should be measured prior to the initiation of study treatment and should be monitored at least weekly, or as defined by the local standard of care, until INR is stable.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment.
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least three months after the last administration of sorafenib.
* Patients may have had a history of other (non-colorectal) malignancies if there is no current evidence of persistent or recurrent disease and they are not undergoing any active therapy (including hormonal).
* Patients should have paraffin-embedded tissue from initial diagnosis or prior colorectal cancer surgery available for molecular analysis.
* Patients must consent to participate in the study and must have signed and dated an IRB-approved consent form conforming to federal and institutional guidelines. Consent must be obtained prior to any study specific procedures.

Exclusion Criteria:

* Prior therapy with a tyrosine kinase inhibitor.
* Age < 18 years
* ECOG Performance Status > 2
* Less than 28 days elapsed from prior radiation therapy, surgery or chemotherapy to the time of registration.
* History of known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* History of clinically significant cardiac disease (severe/unstable angina pectoris, NYHA class III or IV congestive heart failure, symptomatic coronary artery disease) or myocardial infarction, cerebrovascular accident or transient ischemic attack within the last 12 months.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy. Uncontrolled hypertension defined as systolic blood pressure > 140 mmHg or diastolic pressure > 90 mmHg, as measured on 3 consecutive pre-enrollment assessments, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Active clinically serious infection > CTCAE Grade 2.
* Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Pulmonary embolism or any other uncontrolled thromboembolic event within 3 months prior to registration or occurrence of deep vein thrombosis within 4 weeks of registration.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of a clinically significant bleeding diathesis or coagulopathy (without vitamin K antagonist therapy).
* Use of St. John's Wort or rifampin (rifampicin).
* Known or suspected allergy to sorafenib or capecitabine.
* Any condition that impairs patient's ability to swallow whole pills.
* Any known malabsorption problem.
* History of chronic or inflammatory bowel disorders, clinically significant chronic diarrhea refractory to medical management, or unresolved bowel obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-11; Primary Completion 2015-10 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas George, MD, FACP, Principal Investigator — University of Florida
Locations (1):
- UF Health Cancer Center, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 43 Patients were consented and enrolled; however, only 42 were dosed. The one patient that was not dosed was removed due to progression of disease prior to treatment initiation.
Period: Overall Study
Arm/Group | Sorafenib Plus Capecitabine (SorCape)
Started | 42
Completed | 39
Not Completed | 3
Not completed — remain on study | 3

BASELINE CHARACTERISTICS:
Population: Adults with metastatic colorectal cancer who had previously received two or more lines of systemic therapy.
Arm/Group | Sorafenib Plus Capecitabine (SorCape)
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 13
Age, Continuous [Mean (Full Range); unit: years] | 57 [36 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Sorafenib Activity
Description: Determine activity of sorafenib plus capecitabine on progression free survival (PFS) in patients with advanced colorectal cancer. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib Plus Capecitabine (SorCape)
Number analyzed (Participants) | 42
days | 123 [62 to 132]

2. Secondary Outcome: Overall Survival
Description: Evaluate overall survival after treatment.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib Plus Capecitabine (SorCape)
Number analyzed (Participants) | 42
days | 261 [132 to 370]

3. Secondary Outcome: Response Rate
Description: This is the percentage of subjects that achieved either a complete response or a partial response per RECIST 1.1 criteria
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib Plus Capecitabine (SorCape)
Number analyzed (Participants) | 42
percentage of participants | 2.38 [0.06 to 12.57]

4. Secondary Outcome: Response Duration
Description: This is the median response duration (median time from date of a complete or partial response to date of disease progression per RECIST 1.1 criteria) and includes only subjects that achieved either a complete or partial response to treatment per RECIST 1.1 criteria.
Time Frame: up to 12 months
Population: No data are available for this outcome measure since only 1 participant achieved a partial or complete response.
Arm/Group | Sorafenib Plus Capecitabine (SorCape)
Number analyzed (Participants) | 0

5. Secondary Outcome: Toxicity (Percentage of Subjects That Experienced an Adverse Event)
Description: Evaluate acute toxicity of treatment. The toxicity assessments were graded by the NCI CTCAE (Clinical Trial Common Adverse Event) grading system - a global standard for assessments of clinical and laboratory toxicities. All toxicities are scored 1(mild) through 5 (death related to the event) based upon well-defined and reproducible definitions.
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Sorafenib Plus Capecitabine (SorCape)
Number analyzed (Participants) | 42
percentage of participants
  Adverse Events - Any Grade | 100
  Adverse Events - Grade 3 | 74
  Adverse Events - Grade 4 | 2

6. Secondary Outcome: Correlative Tissue Analysis
Description: Exploratory tissue analysis in patients receiving sorafenib plus capecitabine
Time Frame: 6 months
Population: Data were not collected.
Arm/Group | Sorafenib Plus Capecitabine (SorCape)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Sorafenib Plus Capecitabine (SorCape)
Serious Adverse Events (participants affected / at risk) | 13/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib Plus Capecitabine (SorCape) (N=42)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Spleen Disorder (Blood and lymphatic system disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Colonic Obstruction (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Disorders - Other, Bowel Perforation (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
General Disorders and Administration Site Conditions - Other, Anasarca (General disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 2 (3)
Pain (General disorders) | 1 (1)
Hepatobiliary Disorders - Other, Cirrhosis (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Creatinine Increased (Investigations) | 1 (1)
Hyponatremia (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib Plus Capecitabine (SorCape) (N=42)
Abdominal Pain (Gastrointestinal disorders) | 9 (14)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorectal Infection (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 17 (19)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Bloating (Gastrointestinal disorders) | 1 (3)
Blurred Vision (Eye disorders) | 1 (1)
Cardiac Disorders - Other, Ventricular Bigeminy (Cardiac disorders) | 1 (1)
Confusion (Psychiatric disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Creatinine Increasted (Investigations) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Delirium (Psychiatric disorders) | 2 (2)
Delusions (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 16 (30)
Dry Eye (Eye disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 25 (36)
Fever (General disorders) | 1 (3)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Flatulence (Gastrointestinal disorders) | 2 (2)
Flu-Like Symptoms (General disorders) | 4 (4)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Disorders - Other, Gastric Bezoar (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hot Flashes (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 9 (13)
Hypokalemia (Investigations) | 1 (1)
Hyponatremia (Investigations) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Infections and Infestations - Other, Cold Symptoms (Infections and infestations) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Laryngeal Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Localized Edema (General disorders) | 1 (1)
Malaise (General disorders) | 2 (2)
Mucosal Infection (Infections and infestations) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 7 (12)
Musculoskeletal and Connective Tissue Disorder - Other, Muscle Cramps (Musculoskeletal and connective tissue disorders) | 2 (3)
Musculoskeletal and Connective Tissue Disorder - Other, Wrist Sprain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 17 (23)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 2 (8)
Pain (General disorders) | 4 (9)
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 36 (126)
Pelvic Infection (Infections and infestations) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 3 (3)
Personality Change (Psychiatric disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 3 (3)
Platelet Count Decreased (Investigations) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (2)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 4 (4)
Renal Calculi (Renal and urinary disorders) | 1 (2)
Seizure (Nervous system disorders) | 1 (1)
Skin and Subcutaneous Tissue Disorders - Other, Brittle Nails (Skin and subcutaneous tissue disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Splenic Infection (Infections and infestations) | 1 (1)
Syncope (Infections and infestations) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1)
Urine Discoloration (Renal and urinary disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (12)
Weight Loss (Infections and infestations) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes